CLINICAL TRIAL: NCT06179784
Title: Personalising Cognitive Behaviour Therapy for Chronic Primary Pain Using Network Analysis - A Single Case Experimental Design Study With Multiple Baselines
Brief Title: Personalising Psychotherapy for Chronic Primary Pain Using Network Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Julia Glombiewski (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Julia Glombiewski, Clinical professor, Head of department clinical psychology and psychotherapy for adults, University of Kaiserslautern-Landau
Organization: University of Kaiserslautern-Landau (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POINT Pain
Record Dates: First submitted 2023-12-01; First posted 2023-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Primary Pain
Keywords: Chronic Pain; Single Case Experimental Design; Ecological Momentary Assessment; Network analysis; Cognitive Behaviour Therapy
MeSH Terms: conditions — Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to one out of ten treatment modules according to their most relevant pain process. The same module will be used for the whole therapy phase if no adverse effects or long lasting non-response is observed. Only then can the participant be allocated to another treatment module.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Exposure in vivo (Experimental): The goal of the exposure in vivo treatment module is the correction of irrational, fearful beliefs regarding movements, a reduction of avoidance behaviours and hence a facilitation of activity levels. This will be done by carrying out feared, avoided movements and seeking out avoided situations and places. Exemplary units are the development of a movement hierarchy and protocols for exposure exercises.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Relaxation (Experimental): Goal of the relaxation treatment module is the reduction of stress and tension, which will be achieved applying relaxation techniques such as Progressive Muscle Relaxation (PMR), breathing techniques, and imaginary methods.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Activity and Rest (Experimental): The treatment module activity and rest is based on pacing and pursues the goal to balance active and resting phases. For overly active patients, the module will consist of implementing breaks and resting phases, while for overly resting patients the module will consist of graduated activity build-up. Acitivity protocols, plans, and exercises will be used.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Cognitive Coping with Pain (Experimental): Goal of the treatment module cognitive coping with pain is the reduction of rigid, dysfunctional thought patterns by flexibilising them and implement functional thought patterns instead. It includes classical methods such as cognitive restructuring as well as meta-cognitive or defusion techniques.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Attention Control (Experimental): The goal of the treatment module attention control is to enable patients to willingly draw their attention towards other entities as their pain or perceive their pain in a non-judgmental way, thus improve their coping strategies and enhance functioning levels. Exemplary units are the anti-pain diary or the distraction alphabet.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Activating Resources (Experimental): The goal of the activating resources module is relief and a balance between unpleasant perceptions as pain and pleasent experiences. This will be achieved by reactivating lost resources and implementing new ones, e.g. social networks or hobbies. Exemplary units are the positive diary or focusing on healthy bodyparts.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Acceptance (Experimental): Goal of the acceptance module is the flexibilisation of thought patterns by regaining mental resources through givign up inner resistance against the pain. Patients will be supported in developing an accepting attitude towards their suffering using working units like the monster by the wayside or concluding a peace treaty with oneself.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Values and Values-based Action (Experimental): Goal of the treatment module values and values-based action is enhancing satisfaction with life and regaining action control. Patients will learn about their personal values and how they can align their actions with them. Exemplary units are sorting values, a value diary, or looking back on one's life.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Sleep (Experimental): Goal of the treatment module sleep is enhancing the subjective sleep quality and increase the feeling of recovery. Patients will learn about sleep hygiene, stimulus control, and imaginary techniques such as the inner feel-good place.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave
- Selfcompassion (Experimental): Goal of the selfcompassion treatment module is the development of a benevolent, loving, and kind attitude towards oneself and one's suffering in order to enhance wellbeing and feelings of self-worth. Exemplary units are the selfcompassion break, writing a letter to oneself, or changing perspective.
  Interventions: Behavioral: Cognitive Behaviour Therapy including third-wave

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy including third-wave — All treatment modules are based on evaluated treatment manuals and contain methods from Cognitive Behaviour Therapy including methods from the third wave like Acceptance and Commitment Therapy or Mindful Selfcompassion.
  Other Names: Acceptance and Commitment Therapy; Mindful Selfcompassion

SUMMARY:
The goal of this single case experimental design study with multiple baselines is to use network analysis to personalise cognitive behaviour therapy for chronic primary pain (CPP) and base the selection of individual treatment targets and interventions on data to avoid cognitive biases of the clinicians. The main questions it aims to answer are:

* Is the study procedure accepted by and feasible for CPP patients as well as their therapists?
* Does the personalised psychotherapy with databased clinical decisionmaking lead to significant improvement?

Participants will go through several study phases:

* Pretest and informational meeting with study management
* Baseline 1: answering a questionnaire six times a day for 21 days in daily life on their mobilephone (EMA); this data will be used for the calculation of a network for each participant, that in turn will be used to select the treatment target and according treatment intervention as suggested by an algorithmic decisiontool
* Probatory therapy phase: three weekly sessions with therapist; questionnaire three times a week
* Baseline 2: questionnaire three times a week
* Therapy phase: up to ten sessions with therapist; questionnaire three times a week
* Post phase: posttest, two weeks of three weekly assessments, then another 21 days EMA; two monthly booster sessions with therapist
* Follow-up: posttest and meeting with study management

DETAILED DESCRIPTION:
Background and aims:

The treatment of chronic primary pain (CPP) with Cognitive Behaviour Therapy (CBT) is effective, yet effects remain small to moderate. New approaches to the treatment of CPP are needed. They should include an orientation toward processes instead of symptoms and strategies for personalisation. This paradigm shift requests precisce, testable models that allow to link treatment procedures to psychological changes. Unfortunately, current models are rather vague about specific, especially temporal pathways by which its elements interact, or the pathways are not as simplistic as proposed. Therefore, multiple variables and pathways related to the development and persistence of pain-related disabilities should be considered.

One approach to individualisation makes use of repeated measures in the daily lives of patients, which enable the usage of network analysis to investigate interactions between symptoms/processes of a patient. Process-oriented, individualised, network-based therapy for CPP (POINT Pain) combines process-oriented measurements to individualise therapy with network-based analysis approaches for target and treatment selection. We propose the following hypotheses:

1. In line with previous research, we assume that the implementation of POINT Pain is feasible for and accepted by patients as well as therapists. Feasibility and acceptance are indicated by mean ratings of at least 3.5 out of 5 across all items of one scale (each rated on 1-5 Likert scales) on a feedback form developed for this study and by positive comments to open ended questions.
2. Furthermore, we expect POINT Pain to lead to clinically significant improvements as compared to baseline, i.e. decreasing scores in the outcome measures. According to current recommendations, the improvement will be operationalised as effect-size estimated with Hedge's g, the significance with Tau-z.

Procedure:

Before participants are enrolled in the study, they will have two sessions with the study management for diagnostics, pretest, and individualisation of and instructions to the questionnaire.

An ABA'C Multiple Baseline design is chosen to evaluate the effect of individually selected therapy interventions:

Firstly, a baseline assessment (A) is conducted over the period of 21 days six times per day using EMA. In the EMA, a previously validated and piloted questionnaire with items on treatment relevant pain processes is implemented. It contains processes derived from the most prominent psychological models of chronic pain, as there is no overarching theoretical framework adressing the interaction of multi-dimensional pain processes yet. For the EMA, the waking hours of the participants will be divided into six equal time intervals within which the signals for the questionnaires will be randomised (semi randomisation). After completion of phase A, an individual network will be computed.

Secondly, the probatory phase (B) is initiated after completion of phase A. After this phase, an application for psychotherapy is sent to the patient's insurance agency. As much information is already available from phase A, phase B will comprise three sessions. Participants will switch from EMA to SCED assessment in phase B, which means they will answer the same questionnaire as before three times a week, two of which during the week and one on the weekend. The timepoints for the questionnaires will again be semi-randomised during the waking hours of the participants. This procedure stays the same for the remaining phases.

As there is often a natural break between the probatory and the treatment phases due to the psychotherapy application, another baseline (A') is implemented after phase B. The duration of this second baseline will be semi-randomised between one and three weeks.

There are several possibilities for the selection of the most relevant or central variable in a network. The clinical decision regarding treatment target and module will be based on an algorithmic decision-tool which will is programmed based on experts' ratings (see preregistration: https://doi.org/10.17605/OSF.IO/BNFWY). Possible interventions will be limited to a pre-defined intervention pool that was developed based on common therapy manuals for chronic pain. Therapist and supervisor can only rule out the module suggested by the algorithmic decision-tool if there are serious concerns regarding potential harms (e.g. red flags rule out exposure in vivo).

At last, the treatment phase (C) is realised. The selected intervention is carried out until clinically significant improvement is reached or until a maximum of ten sessions has been conducted.

For all assessments using the EMA questionnaire (i.e. phases A to C), the software m-Path (https://m-path.io/landing/) published by KU Leuven will be used.

In addition to the aforementioned assessments, participants will complete traditional outcome measures at three timepoints, i.e. before phase A (pretest), after phase C (posttest), and three months after finishing phase C (follow-up). After phase C, participants will have two more weeks of SCED, after which they will undergo another EMA phase of 21 days with a frequency of six assessments per day in order to calculate a post-therapy network. During this study phase, two monthly booster-sessions with their therapist will take place, but there will not be any further intervention, only monitoring.

The results of the weekly SCED assessments will be analysed in a timely manner and discussed with the participants regularly.

Feasibility and acceptance will be evaluated post-treatment and at follow-up. A feedback form developed for this study will be used for quantitative and qualitative assessment.

Participants:

Patients will be recruited via the waiting list of the university's outpatient clinic, in cooperation with other currently running studies at the same university recruiting chronic pain patients, and via various media (e.g. newspaper articles) and doctors' offices. Study therapists will be recruited in the university's outpatient clinic as well. Inclusion criteria for patients are at least 18 years of age, having access to a smartphone, and the main diagnosis of chronic pain. The diagnosis will be checked using the brief version of the Diagnostic Interview for Mental Disorders (Mini-DIPS). For patients recruited via the waiting list, screening for suitability will take place during the first consultation at the university psychotherapy training centre's outpatient clinic. Suitable participants will be informed about the study and referred if they agree to be contacted. Furthermore, patients that had to be excluded from other currently running studies will be referred if they agreed to be contacted as well.

Analysis:

In the context of SCEDs, each individual can be analysed separately. Especially regarding the qualitative measurements (acceptance, feasibility), it can be assumed that a sample of twelve will lead to a saturation in obtainable answers. Thus, all hypotheses can be answered with a sample of twelve: (1) We can evaluate whether the study procedure is feasible and accepted by patients and therapists, and (2) within SCED clinically significant change can be evaluated per individual. Of course, SCED results will not be generalizable to other individuals.

ELIGIBILITY:
Inclusion Criteria:

* main diagnosis of chronic pain (i.e. pain persists for at least 6 months and is the most prominent/most burdensome symptom)
* subjective impairment/disability (yes-no)
* access to a smartphone compatible with the app mPath

Exclusion Criteria:

* acute hazard due to suicidality, substance abuse, and/or psychosis
* only migraine/headache or migraine/headache are the focus of pain
* analphabetism
* insufficient German knowledge
* current psychotherapy
* current participation in another intervention study
* physical inability to take part in therapy and study sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Ecological Momentary Assessment questionnaire | pre-intervention (two baselines), during intervention (on average 10 weeks + 3 weeks probatory phase), directly after intervention (2 weeks + 21 days)
  Throughout the whole study, the same questionnaire developed and in-evaluation for the use in Ecological Momentary Assessment will be applied. It assesses several therapy-relevant pain processes derived from common psychological models of chronic pain: catastrophising, avoidance, depression (Fear-Avoidance model, Avoidance-Endurance model); thought supression, task persistence, positive affect (Avoidance-Endurance model); acceptance, values (Psychological Flexibility); expectations (Predictive Coding); pain instenisty, pain-related disability (Pain Experience); pain self-efficacy, sleep disturbance, self-compassion. The individual primary outcome will be the most relevant process for each participant according to the network from the first baseline.
Pain Disability Index (PDI) | Pre-intervention, Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  The Pain Disability Index assesses the daily disability caused by pain in seven areas: family/domestic duties, recovery, social activities, work, sexuality, self-care, and life-sustaining activities. It has shown to be a valid instrument, displaying moderate test-retest reliability.
Quebec Back Pain Disability Scale (QBPDS) | Pre-intervention, Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  The Quebec Back Pain Disability Scale will be adapted for chronic pain in general in this study. It assesses disability caused by pain in 20 activities relevant to everyday life. It displays sufficient validity and reliability.

SECONDARY OUTCOMES:
Pain Intensity | Pre-intervention, Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  Pain Intensity will be measured on an 11-point numerical analogue scale over a period of 24 hours.
Short-Form McGill Pain Questionnaire (SF-MPQ) | Pre-intervention, Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  The Short-Form McGill Pain Questionnaire contains of 15 items assessing different pain qualities on a 4-point scale: 11 items assess sensory pain experience, 4 affective pain experience. It also contains a measure of present pain. It is an instrument sensitive enough to detect treatment effects.
German Pain Solutions Questionnaire (PaSol) | Pre-intervention, Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  The German version of the Pain Solutions Questionnaire assesses different coping strategies for pain with 14 items on a 7-point scale: solving pain, meaningfulness of life despite pain, acceptance of the insolubility of pain, and belief in a solution. It displays good reliability and validity and is sensistive for change.
Patient Global Impression of Change (PGIC) | Pre-intervention, Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  One item will be used to assess subjective treatment effects with the Patient Global Impression of Change. It will be answered on a 7-point scale, ranging from "no change" to "very much better".
Pain Self-Efficacy Questionnaire | Pre-intervention, Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  The Pain Self-Efficacy Questionnaire contains on 10 items using a 7-point scale. It was tested regarding comprehensibility and displays high reliability and validity. It also is sensitive to change.
Acceptance and feasibility of study procedures (Feedback form developed for this study) | Post-intervention (directly after intervention), Follow-up (on average three months after intervention)
  Acceptance of the study phases and feasibility will be measured with a feedback form developed for this study, using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- RPTU Kaiserslautern-Landau, Klinische Psychologie und Psychotherapie des Erwachsenenalters, Landau, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elisson LO, Ekberg L. Ifosfamide, doxorubicin, vincristine, and etoposide in small cell lung cancer. Semin Oncol. 1995 Feb;22(1 Suppl 2):15-7. PMID 7846536
- [Background] Williams ACC, Fisher E, Hearn L, Eccleston C. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007407. doi: 10.1002/14651858.CD007407.pub4. PMID 32794606
- [Background] Wright AGC, Woods WC. Personalized Models of Psychopathology. Annu Rev Clin Psychol. 2020 May 7;16:49-74. doi: 10.1146/annurev-clinpsy-102419-125032. Epub 2020 Feb 18. PMID 32070120
- [Background] Vlaeyen JWS, Crombez G. Behavioral Conceptualization and Treatment of Chronic Pain. Annu Rev Clin Psychol. 2020 May 7;16:187-212. doi: 10.1146/annurev-clinpsy-050718-095744. Epub 2019 Dec 10. PMID 31821023
- [Background] Wideman TH, Finan PH, Edwards RR, Quartana PJ, Buenaver LF, Haythornthwaite JA, Smith MT. Increased sensitivity to physical activity among individuals with knee osteoarthritis: relation to pain outcomes, psychological factors, and responses to quantitative sensory testing. Pain. 2014 Apr;155(4):703-711. doi: 10.1016/j.pain.2013.12.028. Epub 2013 Dec 28. PMID 24378879
- [Background] Beeckman M, Simons LE, Hughes S, Loeys T, Goubert L. A Network Analysis of Potential Antecedents and Consequences of Pain-Related Activity Avoidance and Activity Engagement in Adolescents. Pain Med. 2020 Feb 1;21(2):e89-e101. doi: 10.1093/pm/pnz211. PMID 31498397
- [Background] Liew BXW, Ford JJ, Briganti G, Hahne AJ. Understanding how individualised physiotherapy or advice altered different elements of disability for people with low back pain using network analysis. PLoS One. 2022 Feb 10;17(2):e0263574. doi: 10.1371/journal.pone.0263574. eCollection 2022. PMID 35143552
- [Background] Thompson EL, Broadbent J, Fuller-Tyszkiewicz M, Bertino MD, Staiger PK. A Network Analysis of the Links Between Chronic Pain Symptoms and Affective Disorder Symptoms. Int J Behav Med. 2019 Feb;26(1):59-68. doi: 10.1007/s12529-018-9754-8. PMID 30377989
- [Background] Borsboom D. A network theory of mental disorders. World Psychiatry. 2017 Feb;16(1):5-13. doi: 10.1002/wps.20375. PMID 28127906
- [Background] Carlin MT, Costello MS. Statistical Decision-Making Accuracies for Some Overlap- and Distance-based Measures for Single-Case Experimental Designs. Perspect Behav Sci. 2021 Nov 22;45(1):187-207. doi: 10.1007/s40614-021-00317-8. eCollection 2022 Mar. PMID 35342864
- [Background] Morley, S. (2018). Single-case methods in clinical psychology A practical guide (C. M., & C. J. M., Eds.). Routledge.
- [Background] Margraf, J., Cwik, J. C., Suppiger, A., & Schneider, S. (2017). Mini-DIPS Open Access. Diagnostisches Interview bei psychischen Störungen [Short-Form of the Diagnostic Interview for Mental Disorders. Open Access]. https://www.kli.psy.ruhr-uni-bochum.de/dips-interv/klipsy/download/Mini-DIPS%20Open%20Access.pdf
- [Background] Guest, G., Bunce, A., & Johnson, L. (2006). How many interviews are enough?: An experiment with data saturation and variability. Field Methods, 18(1), 59-82. https://doi.org/10.1177/1525822X05279903
- [Background] Turner-Bowker DM, Lamoureux RE, Stokes J, Litcher-Kelly L, Galipeau N, Yaworsky A, Solomon J, Shields AL. Informing a priori Sample Size Estimation in Qualitative Concept Elicitation Interview Studies for Clinical Outcome Assessment Instrument Development. Value Health. 2018 Jul;21(7):839-842. doi: 10.1016/j.jval.2017.11.014. Epub 2018 Mar 7. PMID 30005756
- [Background] Anderson KO, Dowds BN, Pelletz RE, Edwards TW, Peeters-Asdourian C. Development and initial validation of a scale to measure self-efficacy beliefs in patients with chronic pain. Pain. 1995 Oct;63(1):77-83. doi: 10.1016/0304-3959(95)00021-J. PMID 8577493
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Mangels, M., Schwarz, S., Sohr, G., Holme, M., & Rief, W. (2009). Der Fragebogen zur Erfassung der schmerzspezifischen Selbstwirksamkeit (FESS): Eine Adaptation des Pain Self-Efficacy Questionnaire für den deutschen Sprachraum. Diagnostica, 55(2), 84-93. https://doi.org/10.1026/0012-1924.55.2.84
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Tait RC, Chibnall JT, Krause S. The Pain Disability Index: psychometric properties. Pain. 1990 Feb;40(2):171-182. doi: 10.1016/0304-3959(90)90068-O. PMID 2308763
- [Background] Mewes R, Rief W, Stenzel N, Glaesmer H, Martin A, Brahler E. What is "normal" disability? An investigation of disability in the general population. Pain. 2009 Mar;142(1-2):36-41. doi: 10.1016/j.pain.2008.11.007. Epub 2009 Jan 14. PMID 19147292
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Speksnijder CM, Koppenaal T, Knottnerus JA, Spigt M, Staal JB, Terwee CB. Measurement Properties of the Quebec Back Pain Disability Scale in Patients With Nonspecific Low Back Pain: Systematic Review. Phys Ther. 2016 Nov;96(11):1816-1831. doi: 10.2522/ptj.20140478. Epub 2016 May 26. PMID 27231271
- [Background] Sielski R, Glombiewski JA, Rief W, Crombez G, Barke A. Cross-cultural adaptation of the German Pain Solutions Questionnaire: an instrument to measure assimilative and accommodative coping in response to chronic pain. J Pain Res. 2017 Jun 19;10:1437-1446. doi: 10.2147/JPR.S130016. eCollection 2017. PMID 28684921
- [Background] McCracken, L. M. (2005). Contextual cognitive-behavioral therapy for chronic pain. IASP Press.
- [Background] Nicholas, M., Molloy, A., Tonkin, L., & Beeston, L. (2003). Practical and positive ways of adapting to chronic pain Manage your pain. Souvenir press.
- [Background] Kleinstäuber, M., Thomas, P., Witthöft, M., & Hiller, W. (2018). Kognitive Verhaltenstherapie bei medizinisch unerklärten Körperbeschwerden und somatoformen Störungen (2. Aufl.). Springer.
- [Background] Germer CK, Neff KD. Self-compassion in clinical practice. J Clin Psychol. 2013 Aug;69(8):856-67. doi: 10.1002/jclp.22021. Epub 2013 Jun 17. PMID 23775511
- [Background] Germer, C. K., & Neff, K. D. (2019). Mindful Self-Compassion (MSC). In I. Itzvan (Ed.), The handbook of mindfulness-based programs: Every established intervention, from medicine to education (357-367). Routledge.
- [Background] Main, C. J., Keefe, F. J., Jensen, M. P., Vlaeyen, J. W. S., & Vowles, K. E. (2015). Fordyce's Behavioral Methods for Chronic Pain And Illness Republished with Invited Commentaries. IASP Press.
- [Derived] Hofmann VE, Glombiewski JA, Kininger F, Scholten S. How to personalise cognitive-behavioural therapy for chronic primary pain using network analysis: study protocol for a single-case experimental design with multiple baselines. BMJ Open. 2024 Dec 3;14(12):e089319. doi: 10.1136/bmjopen-2024-089319. PMID 39627123
- See also: Preregistration of the algorithmic decision-tool — https://doi.org/10.17605/OSF.IO/BNFWY
- See also: Preregistration of the EMA questionnaire development — https://doi.org/10.17605/OSF.IO/S4RMN
- See also: Assessment app mPath — https://m-path.io/landing/